CLINICAL TRIAL: NCT05245903
Title: Passive Sensor Identification of Digital Biomarkers to Assess Effects of Orally Administered Nicotinamide Riboside on Bioenergetic Metabolism, Oxidative Stress, and Cognition in Mild Cognitive Impairment and Mild Alzheimer's Dementia
Brief Title: Passive Sensor Identification of Digital Biomarkers to Assess Effects of Orally Administered Nicotinamide Riboside
Acronym: Emerald-NRAD
Status: Recruiting | Type: Observational
Sponsor: Mclean Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Ipsit Vihang Vahia, Associate Chief of Geriatric Psychiatry, Mclean Hospital
Other Study IDs: 2021P003275
Record Dates: First submitted 2021-12-21; First posted 2022-02-18 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Alzheimer Disease; Dementia Alzheimers; Dementia; Cognitive Impairment; Mild Cognitive Impairment; Neurodegenerative Diseases; Neurocognitive Disorders; Neurocognitive Dysfunction; Cognitive Dysfunction; Mental Disorder
Keywords: Passive sensing; Digital phenotyping; Alzheimer's Dementia; Mild Cognitive Impairment; Digital biomarker
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction; Neurodegenerative Diseases; Neurocognitive Disorders; Cognition Disorders; Mental Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Parent Study Participants: The single group in this study will consist of individuals enrolled in the parent study (ClinicalTrials.gov identifier NCT04430517). We aim to enroll approximately 40 individuals aged 18 -89 (inclusive) with either MCI or mild AD who will have the Emerald device deployed in their home for up to 12 weeks, spanning the time of approval of parent study screening and formal study enrollment.
  Interventions: Device: Emerald Device Monitoring

INTERVENTIONS:
Device: Emerald Device Monitoring — The study participants will have the Emerald device deployed in their home for up to 12 weeks as they participate in the parent study (ClinicalTrials.gov identifier NCT04430517). The device will be deployed in the bedroom of each subject to capture behavior continuously. The Emerald device is a radio-wave sensor that will use signal processing and machine learning algorithms to track the gait, movement, respiration, and sleep of these subjects via low-powered radio signals. Reflections of the radio signals are processed using algorithms to convert them into movement data, sleep stages, and key sleep parameters. These data will supplement bioenergetic, imaging, and biochemical data with digital biomarkers and phenotyping using this device.

SUMMARY:
This project's main goal is to use state-of-the-art passive sensing techniques to identify digital biomarkers that relate to bioenergetic changes in the brain due to nicotinamide riboside supplementation in those with mild cognitive impairment and mild Alzheimer's dementia.

DETAILED DESCRIPTION:
The investigators will conduct a prospective, single-arm, non-interventional study using the Emerald device to monitor the behavior of individuals enrolled in the parent study (ClinicalTrials.gov identifier NCT04430517). Investigators aim to enroll approximately 40 individuals aged 18 -89 (inclusive) with either MCI or mild AD who will have Emerald deployed in their home for up to 12 weeks, spanning the time of approval of parent study screening and formal study enrollment. The Emerald device is a radio-wave sensor that uses signal processing and machine learning algorithms to track the gait, movement, respiration, and sleep of subjects without physical contact or effort by the user, i.e. it neither requires the subject to wear a sensor nor record any data. Emerald works by transmitting low-powered radio signals, 1000x less than Wi-Fi, that reflect off of the subject and return back to the device. If the user moves their arm or leg, or their chest expands and contracts from breathing, that movement changes how the signal reflects off of their body. Emerald records these reflections and processes them using algorithms that convert the radio signals into movement data, breathing rate, sleep stages (Awake, Light, Deep and REM), and key sleep parameters. The device will be deployed in the bedroom of each subject to capture behavior continuously.

ELIGIBILITY:
Inclusion Criteria:

* Ability of the participant and/or his/her legally authorized representative to understand the purpose and risks of the study, to provide signed and dated informed consent, and to authorize the use of confidential health information.
* Ability to speak and read fluently in English
* 18-89 years old (inclusive)
* Normal or corrected to normal hearing and vision
* Meet clinical diagnostic criteria for MCI or Mild AD, according to the criteria outlined above
* Study partner available for duration of trial participation
* At least one copy of the APOE ε4 allele
* An aggregate risk score > 4 according to the risk analysis method developed by Sabbagh et al. (2017)
* For individuals who are taking niacin (or a vitamin supplement with niacin) of >200mg, the completion of a two-week wash-out period

Exclusion Criteria:

* Current serious or unstable medical or neurological condition that could affect cognitive functioning, as determined by study clinician
* Clinically unstable mood or anxiety disorder within 6 months prior to screening, as determined by study clinician
* Lifetime history of psychotic disorder (i.e. Schizophrenia, Schizoaffective Disorder), as determined by study clinician
* Diagnosis of a mitochondrial disorder
* Any MRI safety contraindications
* History of drug hypersensitivity or intolerance to NR
* Transient ischemic attack or stroke within 1 year prior to screening
* History of alcohol or substance abuse within prior year, as determined by study clinician and urine toxicology screen
* History of head injury rated as moderate or worse, per DSM-5 criteria
* History of seizure within prior 10 years
* Current use of medication with known adverse effects on cognition (benzodiazepines, barbiturates, opiate analgesics, first generation antipsychotic medication, anticholinergics, sedating antihistamines, tricyclic anti-depressants)
* Change in dose of any psychiatric medications within 4 weeks of screening visit
* Prior use of L-DOPA, any anti-Parkinsonian medication, or prior treatment with anti-amyloid immunotherapy
* Current use of putative mitochondrial enhancers or antioxidants (e.g. carnitine, creatine, Co-Q10, N-acetyl cysteine, pramipexole)
* Initiation of treatment or change in dosing of acetylcholinesterase inhibitors (AChEIs) and memantine within 4 weeks of screening
* Prior use of prescription narcotics 4 weeks before screening
* Female subjects who are pregnant or breastfeeding
* The current use of niacin (or a vitamin supplement with niacin) >200mg within the last two weeks prior to study visit

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the existing pool of study subjects for the parent study (MGB IRB protocol #2020P001652, ClinicalTrials.gov identifier NCT04430517). Participation in this supplemental portion of the parent study will be elective for study subjects. Separate informed consent for the installation of the Emerald device will be used, and recruitment for this study will run concurrently with the parent project (IRB protocol #2020P001652, ClinicalTrials.gov identifier NCT04430517). All consented individuals will be targeted for supplemental recruitment for this project.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Sleep efficiency | Week 0 to week 12 of parent study (ClinicalTrials.gov identifier NCT04430517)
  Sleep efficiency will be measured by the Emerald as a ratio of the total sleep time to the time in bed supplemented by tracking participants' wake after sleep onset (WASO), sleep stages (light, deep, REM), sleep latency, and number of awakenings per night.
Longitudinal time series of gait speed measurements | Week 0 to week 12 of parent study (ClinicalTrials.gov identifier NCT04430517)
  Gait speed will be measured by the Emerald device and developed into a longitudinal time series of gait speed (meters per second) throughout the 12-week study.
Diurnal rhythm | Week 0 to week 12 of parent study (ClinicalTrials.gov identifier NCT04430517)
  The diurnal rhythms of study participants will be extracted by using the Emerald device to track patients' spatial location within their living environment and quantifying levels and patterns of motion. This will serve as a marker of psychomotor activity.

CONTACTS AND LOCATIONS:
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No